CLINICAL TRIAL: NCT07019558
Title: Ophthalmological Disorders in Dominant Spinal-cerebellar Ataxias
Acronym: AO-SCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL24_0301
Record Dates: First submitted 2025-05-28; First posted 2025-06-13 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Spinocerebellar Ataxia
Keywords: spinocerebellar ataxias; ophtalmology; neurology
MeSH Terms: conditions — Spinocerebellar Ataxias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): * Symptomatic subjects with SCA1, SCA2 or SCA3, symptomatic subjects with SCA27B.
  * Presymptomatic subjects carrying the mutation for SCA1, SCA2 and SCA3.
  Interventions: Other: Neurological assessment; Diagnostic Test: Ophthalmological assessment

INTERVENTIONS:
Other: Neurological assessment — Collect retrospective and current clinical data and assess motor impairment
Diagnostic Test: Ophthalmological assessment — Ophthalmological assessment of possible optic nerve or retinal damage.

SUMMARY:
Spinocerebellar ataxias (SCA) are rare genetic neurological disorders. The most common forms are SCA1, SCA2 and SCA3. Another more recently identified cause of ataxia is SCA27B.

These are progressive, incapacitating pathologies, with adult onset (generally between 30 and 60 years of age) and progressive involvement. They are characterized by gait instability (ataxia), coordination disorders (dysmetria) and speech disorders (dysarthria). A complex disorder may also be present, with impaired ocular motility, double vision (diplopia) and difficulties with eye movements (ophthalmoplegia).

In clinical practice, investigators have observed patients with advanced forms of SCA1 or SCA3 reporting a progressive decline in visual acuity. Other recent scientific observations confirm the possible presence of additional ophthalmological damage to the retina or optic nerve in SCA1, SCA2 and SCA3 pathologies.

This study is a cross-sectional study, including subjects with SCA1, SCA2 and SCA3 at different stages of the disease, including the presymptomatic stage, with a complete and systematic study of visual damage.

The same study will be applied to subjects with SCA27B in order to study the presence or absence of visual impairment, and possibly compare it with those of patients with polyglutamine-expanded SCA.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80,
* Presence of pathological expansion in ATXN1 (> or equal to 39 CAG), ATXN2 (> or equal to 33 CAG) or ATXN3 (> or equal to 45 CAG) genes, responsible respectively for SCA1, SCA2 or SCA3 or a pathological expansion (>250 GAA) in the FGF14 gene responsible for SCA27B pathology,
* Sujet symptomatic (SARA greater than or equal to 4) or presymptomatic (SARA < 4).

Exclusion Criteria:

* Study-specific criteria:

  * Subjects with systemic or ophthalmological disease that could affect the retina, impair fundus examination (severe cataract, severe/decompensated diabetes), or cause visual acuity below 20/40, intraocular pressure > 20 mmHg, "cup to disc" ratio > 0. 5, or severe refractive errors
  * Subjects with extremely severe neurological impairment, with a significant impact on the ability to perform most ophthalmological examinations; for example in patients for whom sitting, even with back support and cannot be maintained. The possibility of including subjects with a severe form will be evaluated on a case-by-case basis, according to the opinion of the principal investigator and the ophthalmologist.
* General exclusion criteria relating to regulations:

  * Failure to obtain consent (adults, non-emancipated minors, persons not in a position to give consent, research carried out in emergency situations, etc.),
  * Participants who have reached the maximum amount of compensation for their participation inresearch,
  * Non-affiliation with a social security scheme,
  * Persons placed under court protection,
  * Person taking part in research.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Percentage (%) of patients with SCA1, SCA2, or SCA3 showing abnormalities for each ophthalmological examination performed. | 1 day
  * Visual Acuity Assessment: Significant reduction in visual acuity (<5/10) unexplained by other causes (such as age or other diseases).
  * Color Vision: Normal or pathological, with description of the axis
  * Fundus Examination: Normal or pathological (presence of retinopathy or optic nerve atrophy).
  * Optical Coherence Tomography (OCT): Evaluation of retinal nerve fiber layer (RNFL) and macular thickness (at 3 mm and 6 mm from the center), including retinal thickness, ganglion cell layer thickness, and the status of the ellipsoid zone. These thickness measurements are quantified according to age-adjusted normative database values.
  * Visual Evoked Potentials (VEP): Normal or pathological; if pathological, characterized by prolonged conduction times and/or reduced amplitude.
  * Electroretinogram (ERG): Normal or pathological; if pathological, defined by alteration (>2 standard deviations) in the amplitude or latency of a- or b-waves under photopic or scotopic conditions

SECONDARY OUTCOMES:
Percentage (%) of subjects showing abnormalities for each ophthalmological examination performed | 1 day
  Percentage (%) of subjects showing abnormalities for each ophthalmological examination performed to compare disorder across the three different types of SCA.
Severity of clinical impairment assessed by the SARA score (Scale for the Assessment and Rating of Ataxia) and the associated disability scale. | 1 day
  Severity of clinical impairment assessed by the SARA score (Scale for the Assessment and Rating of Ataxia) and the associated disability scale to correlate ophthalmological abnormalities. The SARA is a tool for assessing ataxia. It has eight categories with accumulative score ranging from 0 (no ataxia) to 40 (most severe ataxia) where higher scores indicate worse clinical impairment.
Disease duration: number of years between the estimated symptom onset and the time of study inclusion. | Day 1
  Disease duration: number of years between the estimated symptom onset and the time of study inclusion to assess whether this disorder is early and already present at a presymptomatic stage

OTHER OUTCOMES:
Percentage (%) of patients with SCA27B showing abnormalities for each ophthalmological examination performed. | 1 day
  * Visual Acuity Assessment: Significant reduction in visual acuity (<5/10) unexplained by other causes (such as age or other diseases).
  * Color Vision: Normal or pathological, with description of the axis
  * Fundus Examination: Normal or pathological (presence of retinopathy or optic nerve atrophy).
  * Optical Coherence Tomography (OCT): Evaluation of retinal nerve fiber layer (RNFL) and macular thickness (at 3 mm and 6 mm from the center), including retinal thickness, ganglion cell layer thickness, and the status of the ellipsoid zone. These thickness measurements are quantified according to age-adjusted normative database values.
  * Visual Evoked Potentials (VEP): Normal or pathological; if pathological, characterized by prolonged conduction times and/or reduced amplitude.
  * Electroretinogram (ERG): Normal or pathological; if pathological, defined by alteration (>2 standard deviations) in the amplitude or latency of a- or b-waves under photopic or scotopic conditions

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier - Hôpital Gui de Chauliac, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: Undecided